CLINICAL TRIAL: NCT01230125
Title: Study to Assess the Efficacy and Safety of Mapracorat Ophthalmic Suspension, 3% in Subjects for the Treatment of Ocular Inflammation Following Cataract Surgery
Brief Title: Mapracorat Ophthalmic Suspension for the Treatment of Ocular Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 663
Record Dates: First submitted 2010-10-25; First posted 2010-10-28 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Cataract
Keywords: Inflammation; Pain; Ocular surgery
MeSH Terms: conditions — Cataract; Inflammation; Pain | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mapracorat (Experimental): Ophthalmic suspension 3%
  Interventions: Drug: Mapracorat
- Vehicle (Placebo Comparator): Vehicle of mapracorat ophthalmic suspension
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Mapracorat — Instill study medication into study eye per dosing instructions for 14 days
  Other Names: BOL-303242-X
  Arms: Mapracorat
Drug: Vehicle — Instill study medication into the study eye per dosing instructions for 14 days
  Arms: Vehicle

SUMMARY:
The objective of this clinical study is to compare the safety and efficacy of Mapracorat Ophthalmic Suspension, 3% to vehicle for the treatment of postoperative inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are candidates for routine, uncomplicated cataract surgery
* Participants who, in the Investigator's opinion, have potential postoperative pinhole Snellen visual acuity (VA) of at least 20/200 in the study eye.
* Participants must be willing to wait to undergo cataract surgery on the fellow eye until after the study has been completed.

Exclusion Criteria:

* Participants who are expected to require concurrent ocular therapy (either eye) with nonsteroidal anti-inflammatory drugs (NSAIDs), mast cell stabilizers, antihistamines, or decongestants.
* Participants who are expected to require treatment with any systemic or ocular (either eye) corticosteroids or glucocorticoids.
* Participants who are expected to require concurrent ocular therapy with immunosuppressants (eg, Restasis).
* Participants who have known hypersensitivity or contraindication to the study drug(s) or their components.
* Participants participating in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mapracorat | Vehicle
Started | 207 | 104
Completed | 134 | 54
Not Completed | 73 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mapracorat | Vehicle | Total
Number analyzed (Participants) | 207 | 104 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.75) | 69.0 (7.53) | 69.1 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 58 | 167
  Male | 98 | 46 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells.
Description: Anterior chamber (AC) cells were assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 207 | 104
Participants | 32 | 12

2. Primary Outcome: Percentage of Participants With Grade 0 Pain
Description: Ocular pain was defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. The scores ranged from 0=None to 5=Severe, were higher scores indicated worse pain.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 207 | 104
Participants | 130 | 57

3. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Flare.
Description: A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens will be performed without pupil dilation. Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). The grades for flare were 0=None to 4=Very Severe effect.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mapracorat | Vehicle
Number analyzed (Participants) | 207 | 104
Participants | 90 | 30

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | Mapracorat | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/207 | 0/104
Other Adverse Events (participants affected / at risk) | 14/207 | 17/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mapracorat (N=207) | Vehicle (N=104)
Cystoid macular edema (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mapracorat (N=207) | Vehicle (N=104)
Eye pain (Eye disorders) | 9 | 10
Corneal edema (Eye disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.